CLINICAL TRIAL: NCT02923336
Title: Evaluation of Gastrointestinal Transite in Cirrhotic Patient Pre and Post Treatment With Non Selective Betablockers (Propanolol)
Brief Title: Evaluation of Gastrointestinal Transit Pre and Pos Treatment With Non Selective Betablocker in a Population of Cirrhotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ALDO TORRE DELGADILLO (Other)
Responsible Party: Sponsor-Investigator, ALDO TORRE DELGADILLO, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GAS-1068-13/15-1
Record Dates: First submitted 2016-10-02; First posted 2016-10-04 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; variceal bleeding; non selective beta blockers
MeSH Terms: conditions — Liver Cirrhosis | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smart pill (Other): Single group, before and after, the same group is going to be its own control
  Interventions: Drug: non selective beta blocker

INTERVENTIONS:
Drug: non selective beta blocker — the patient is going to receive a device called "smart pill" before the beginning of treatment with propranolol, after the evaluation with the smart pill device, they are goning to take propranolol (dose of propranolol 80 mg per day) for 4 weeks,finally they will receive another smart pill to evaluate the second gastrointestinal transit time
  Other Names: propranolol

SUMMARY:
The purpose of this study is to evaluate the influence of non betablockers in gastrointestinal motility (transit time) in patients with liver cirrhosis.

DETAILED DESCRIPTION:
There is some evidence that cirrhotic patients have increased gastrointestinal transit time, this issue may favor bacterial owergrowth, and consequently bacterial translocation. Translocation of bacterias and its products are linked to vascular and hemodynamics alterations that produce descompensation on the disease. There is evidence , in animal models , that the use of beta blockers favors the gastrointestinal movement; decompensated cirrhotics had significantly longer small bowel transit time as compared with compensated cirrhotics, there have described that this alteration is related to de cirrhosis severity as assessed by Child Pugh score. The purpose of this study is to evaluate the gastrointestinal transit time before and after treatment of non selective betablockers, we are going to evaluate the gastrointestinal time before and after of 4 weeks of non selectivebetablocker treatment, in decompensated cirrhotics. The gastrointestinal time is going to be evaluate by the ingestion of a device known as "smart pill", that allow ambulatory monitoring of gastrointestinal transit.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any ethiology
* Child Pugh A, B, C without beta-blocker treatment previously (min. 1 month without treatment)
* Patients with previous variceal bleeding (with liver cirrhosis) * Patients with ascites or bacterial spontaneous peritonitis

Exclusion Criteria:

* Variceal disease without cirrhosis
* Cirrhotics patients that use antibiotics, prebiotics and probiotics during the study period and one month previously
* Patients under immunosuppressor treatment
* Patients with portal thrombosis
* Patients with Sd. Budd-Chiari or cava/suprahepatic thrombosis
* Patients with active infection process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-01 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal transit time before and after treatment with no selective betablocker | 4 weeks of maximum non betablocker dose
  gastrointestinal time evaluated by a device called Smart pill
Evaluatiuon of genes of tight junctions proteins before and after treatment with no selective betablocker | 4 weeks of maximum non betablocker dose
  gene expression of tight junctions proteins in duodenal and gastric epithelium

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas Y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Chander Roland B, Garcia-Tsao G, Ciarleglio MM, Deng Y, Sheth A. Decompensated cirrhotics have slower intestinal transit times as compared with compensated cirrhotics and healthy controls. J Clin Gastroenterol. 2013 Nov-Dec;47(10):888-93. doi: 10.1097/MCG.0b013e31829006bb. PMID 23632359